CLINICAL TRIAL: NCT04327219
Title: Prospective Dietary Therapy Using Crohn's Disease Exclusion Diet ("CDED") for Ileal Pouch Anal Anastomosis ("IPAA") Patients With Endoscopic Deterioration or Clinically Suspected Pouchitis
Brief Title: Prospective Dietary Therapy Using Crohn's Disease Exclusion Diet for Ileal Pouch Anal Anastomosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, PI, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-0637-19-CTIL
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Pouchitis; Crhon's Disease Like of the Pouch
Keywords: pouchitis; crohn's disease of the pouch; crohn's disease exclusion diet; CDED; ileal pouch anal anastomosis; IPAA
MeSH Terms: conditions — Pouchitis

STUDY DESIGN:
Intervention Model Description: 1. Twenty patients, at 0-3 months post ileostomy closure will be enrolled for the study. Patients will be randomized to receive the CDED or standard diet at a ratio of 1:1
  2. Fourty two adults with a diagnosis of acute exacerbation of pouchitis will be included in the study. Participants will be randomised to receive the CDED or standard diet at a ratio of 1:1.
  Upon initiation of the patient recruitment, 15 pouchitis patients will be treated with the study diet (modified CDED) for 24 weeks per treatment protocol as a pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDED diet (Experimental): The CDED will be divided into 3 stages: 0-6 weeks- induction phase (phase 1), weeks 7-12 step-down phase (phase 2), week 13 -24 maintenance phase (phase 3). During these weeks the diet is structured and contains a list of allowed/disallowed foods, and mandatory foods with specific daily/weekly amounts. Patients will be asked to progress with the diet if they respond to the diet clinically. Patients who do not improve, but show a clinicaly significant trend in symptoms, may be asked to prolong a dietary phase until reaching clinical reaction.
  Interventions: Other: CDED diet
- standard diet (No Intervention): The control standard diet will be personally tailored for nutritional needs according to patient's daily recommended intake (DRI) for calories and protein intake (25kcal/kg and 0.8-1gr/kg per day respectivlly), and will follow the clinical guidelines for dietary therapy of patients with IBD.

INTERVENTIONS:
Other: CDED diet — examine the microbial, mucosal and immunological changes of the pouch during one year post IPAA, and examine the impact of the CDED on disease activity and dysbiosis in adults suffering from active pouchitis.
  Arms: CDED diet

SUMMARY:
Restorative proctocolectomy with ileal pouch-anal anastomosis (IPAA) is the surgical treatment of choice for patients with ulcerative colitis (UC) who require surgery. Inflammation of the ileal pouch (pouchitis) occurs in up to 60% of pouch patients.

Although, pouchitis patients are former UC patients, the disease occurs in the small intestine, similarly to Crohn's disease (CD). Further, the disease can be clinically similar to CD, involving the proximal gastro-intestinal tract and causing strictures, fistula, or perianal disease.

The Crohn's Disease Exclusion Diet (CDED) reduces exposure to all the components identified in rodent models as well as two components that are highly suspect but have not been investigated in models. The diet also provides dietary components that may favor species (especially SCFA producers) which appear to be deficient in CD.

The investigator therefore aims to examine the microbial, mucosal and immunological changes of the pouch during one year post IPAA, and examine the impact of the CDED on disease activity and dysbiosis in a cohort of adults suffering from active pouchitis.

DETAILED DESCRIPTION:
Hypothesis (es) and Aims:

1. The investigator aims to evaluate the natural development of the pouch microenvironment among post-IPAA patients over one year of follow-up, and associate dietary intake with shaping the pouch microbiome composition, metabolic activity, proteolytic activity and with development of pouchitis.

   The investigator hypothesizes that the different dietary pattern of post-IPAA patients will be associated with different pouch microenvironments, and with the development of pouchitis.
2. The investigator aims to measure the effect of the CDED on shaping the pouch microenvironment among post-IPAA patients over one year of follow-up, compared with a control standard diet. The investigator further aims to assess if the CDED is an effective mean of prevention of pouchitis in post-IPAA patients.

   The investigator hypothesizes that adherence to the CDED post-IPAA will positively effect the pouch microbiome composition, metabolic activity and proteolytic activity, and be an efficient means to maintain surgical remission in pouch patients, compared with a control standard diet.
3. The investigator aims to evaluate the effect of the CDED on acute pouchitis activity compared with a control-standard diet.

   The investigator hypothesizes that the CDED will induce clinical, biological and endoscopic remission in pouchitis patients, and that remission will be maintained through 24 weeks. Results are expected to show superiority over a standard diet for clinical remission in pouchitis patients.
4. The investigator aims to examine whether changes in circadian rhythm are associated with improvement in clinical and biological disease activity.

Study plan:

1. POST IPAA SURGERY PATIENTS:

   1.1 Twenty patients, at 0-3 months post ileostomy closure will be enrolled for the study. Patients will be randomized to receive the CDED or standard diet at a ratio of 1:1. Patients will undergo 5 clinic visits for dietary education and guidance at baseline, weeks 3, 6, 12 and 24 in which they would be closely monitored for dietary adherence, physician assessment of disease ativity, patient reported outcomes (PROMS) and quality of life. Patient followup under the CDED maintenance phase, including data collection will continue every 8 weeks up to 52 weeks.

   1.2 Pouchoscopy will be performed at baseline (unless preformed within 2 months of inclusion), week 12, week 24 and week 52, to assess pouchitis activity and to retrieve mucosal samples for histology, mucosal adherent bacteria assessment, and RNA extraction 1.3 Screening: At baseline, inclusion and exclusion criteria will be evaluated, informed consent obtained and participants asked to provide stool, urine and blood samples, undergo anthropometric evaluation, and fill in lifestyle, quality of life and nutritional questionnaires.

   Baseline pouchoscopy will include validation of endoscopic inclusion criteria and sampling of intestinal tissue.

   Patients will be randomized to undergo the CDED or receive a standard diet personally tailored for patient's nutritional needs and symptoms by a trained dietitian.

   1.4 Follow-up Patients will be evaluated for a disease activity index (mPDAI), CBC, CRP, calprotectin, albumin and weight at each of the visits (baseline, week 3, week 6, week 12, week 24 and week 52). Biological samples will be analyzed and preserved for future analysis at -80 at each visit.

   Dietary compliance will be assessed by a modified MARS questionnaire at each visit and by dieticians using a 3 days food diary at four time points (week 3 , 6, 12 and 24), and two telephone calls one week after each change at weeks 1 and 7.

   All patients will undergo a pouchoscopy at the end of 12 and 24 weeks of the diet for evaluation of disease activity and tissue sample collection.

   After week 24, patients who do not respond to treatment at either arm, will be defined as treatment failures. Those who do respond and who achieve steroid free clinical remission, will be instructed to continue with the maintenance diet until week 52 of the study followup.
2. study plan: 2.1 Fourty two adults with a diagnosis of acute exacerbation of pouchitis will be included in the study. Participants will be randomized to receive the CDED or standard diet at a ratio of 1:1. Patients will undergo 5 clinic visits for dietary education and guidance at baseline, weeks 3, 6, 12 ans 24 in which they would be closely monitored for dietary adherence, physician assessment of disease activity, patient reported outcomes (PROMS) and quality of life.

After 6 weeks of CDED phase 1, patients will be clinically evaluated to define clinical response as reduction in clinical PDAI>1 point. Patients receiving the standard diet who do not achieve clinical remission at week 6 will be able to be re-allocated to the CDED arm per protocol. Patients who do achieve remission will continue with their tailored diet until week 24.

Pouchoscopy will be performed at baseline (unless preformed within 2 months of inclusion), week 12 and week 24 to assess pouchitis activity and to retrieve mucosal samples for histology, mucosal adherent bacteria assessment, and RNA extraction 2.2 Follow-up: Patients will be evaluated for a disease activity index (mPDAI), CBC, CRP, calprotectin, albumin and weight at each of 5 visits (baseline, week 3, week 6, week 12, and week 24). Biological samples will be analyzed and preserved for future analysis at -80 at each visit.

Dietary compliance will be assessed by a modified MARS questionnaire at each visit and by dieticians using a 3 days food diary at four time points (week 3 , 6, 12 and 24), and two telephone calls one week after each change at weeks 1 and 7.

All patients will undergo a pouchoscopy at the end of 12 and 24 weeks of the diet for evaluation of disease activity and tissue sample collection.

ELIGIBILITY:
Inclusion Criteria:

1. Post-IPAA for ulcerative colitis ≤3 months post-opp OR post -IPAA for UC 1.1 Active pouchitis defined as: 1.1.1 ≥5 points modified Pouch disease activity index (mPDAI), and one of the following: 1.1.2 Pouchoscopy demonstrating lesions in the ileum/jejunum/afferent pouch loop of the pouch, clinical PDAI>2 points 1.1.3 MR/CTEnterography with evidence of inflammation of the pouch 1.1.4 Fecal calprotectin>250 µg/gr
2. Lack of obstructive symptomes for 8 weeks
3. Stable medications and doses:

   3.1 Immunomodulatory and biologics at least 8 weeks 3.2 Mesalamine at least 4 weeks 3.3 Medical cannabis at least 2 weeks 3.4 Budesonide dependent allowed if patients are active and budesonide dose is ≤6 mg, VIVOMIX probiotics allowed). Use of Antibiotics / Budesonide <6 mg at baseline*.

   *Patients treated with steroids or antibiotics at baseline will be included in the study and be allowed to continue the study if they treated with a stable dose throughout at least 4 weeks. After 4 weeks if the trial, if they present clinical improvement, according to the judgment of the study physician, dose may be gradually reduced for the remaining trial without exclusion.
4. Informed consent and ability to complete the study protocol.

Exclusion Criteria:

1. Pregnancy
2. Use of systemic steroids / Budesonide >6 mg at baseline.
3. Currently active systemic diseases such as spondylo-arthropathies, collagen vascular disease, renal failure, hepatitis or heart disease
4. Positive Stool culture, stool parasites or clostridium difficile toxin or alternative C- Difficile test.
5. Evidence of bowel stricture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
steroid free clinical remission | week 6
  defined as Clinical pouchitis disease activity index ("cPDAI" ranges between 0-6 where highest is the worst and lowest is best clinically) sub score≤2 for pouchitis patients

SECONDARY OUTCOMES:
Steroid free clinical remission | week 12
  defined as Clinical pouchitis disease activity index ("cPDAI" ranges between 0-6 where highest is the worst and lowest is best clinically) sub score≤2
Maintenance of clinical remission | week 24
  defined as Clinical pouchitis disease activity index ("cPDAI" ranges between 0-6 where highest is the worst and lowest is best clinically) sub score≤2
clinical and endoscopic remission | week 12
  defined as modified pouchitis disease activity index ("mPDAI" ranges between 0-12 where highest is the worst and lowest is best clinically) sub score<5
clinical and endoscopic remission | week 24
  defined as modified pouchitis disease activity index ("mPDAI" ranges between 0-12 where highest is the worst and lowest is best clinically) sub score<5
Clinical response | week 6
  reduction in Clinical pouchitis disease activity index ("cPDAI" ranges between 0-6 where highest is the worst and lowest is best clinically) ≥1
Clinical response | week 12
  reduction in Clinical pouchitis disease activity index ("cPDAI" ranges between 0-6 where highest is the worst and lowest is best clinically) ≥1
Pouchitis remission | week 12
  defined as pouchitis disease activity index ("PDAI" ranges between 0-18 where highest is the worst and lowest is best clinically) <7 points
Pouchitis remission | week 24
  defined as pouchitis disease activity index ("PDAI" ranges between 0-18 where highest is the worst and lowest is best clinically) <7 points
Clinically significant change in mean CRP | week 6
  normalization (CRP ≤5mg/l) of CRP or reduction in CRP of ≥10 mg/l
Clinically significant change in mean CRP | week 12
  normalization (CRP ≤5mg/l) of CRP or reduction in CRP of ≥10 mg/l
Clinically significant change in mean CRP | week 24
  normalization (CRP ≤5mg/l) of CRP or reduction in CRP of ≥10 mg/l
Clinically significant change in mean fecal calprotectin | week 6
  normalization (≤150 mg/g) in calprotectin or reduction in calprotectin of ≥150mg/gr
Clinically significant change in mean fecal calprotectin | week 12
  normalization (≤150 mg/g) in calprotectin or reduction in calprotectin of ≥150mg/gr
Clinically significant change in mean fecal calprotectin | week 24
  normalization (≤150 mg/g) in calprotectin or reduction in calprotectin of ≥150mg/gr

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel